CLINICAL TRIAL: NCT04919083
Title: Effects of a Multimodal Program of Therapeutic Exercise and Functional Recovery With Follow-up in the Elderly After Hip Fracture Surgery Using a Digital Application. Observational Study.
Brief Title: Exercise Program and Follow-up in the Elderly After Hip Fracture Surgery Using a Digital Application.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zamar Fisioterapia (Other)
Collaborators: Hospital San Juan de Dios, Spain (Other); Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Joaquín Zambrano-Martín, Principal Investigator, Zamar Fisioterapia
Other Study IDs: P_2020_007_v1
Record Dates: First submitted 2021-05-20; First posted 2021-06-09 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Hip Fractures
Keywords: Hip fractures; Physiotherapy; Functional capacity; Frail elderly
MeSH Terms: conditions — Hip Fractures | interventions — Recovery of Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-exposed cohort (protective factor): Group of patients operated on during the year 2021 in San Juan de Dios Hospital for hip fracture and to which the new programme implementing functional recovery and therapeutic exercise will be applied with follow-up for one year. The implementation of a functional recovery plan and subsequent follow-up is considered a protective factor in relation to the loss of functionality.
  Interventions: Other: Program of Therapeutic Exercise and Functional Recovery
- Exposed cohort (retrospective): Complete cohort of patients operated on during the year 2020 in San Juan de Dios Hospital for hip fracture and to whom no specific functional recovery plan was applied.
  Interventions: Other: Standardised nursing care plan

INTERVENTIONS:
Other: Program of Therapeutic Exercise and Functional Recovery — Specific hip fracture recovery programme,restoring the mobility, strength and balance of the operated patient, in order to facilitate the return to a functional state as close as possible to the state prior to surgery and in the shortest possible time, as detailed in Annex VIII. This programme is part of the standard treatment protocol implemented since January 2021 by the Orthogeriatrics Unit of the San Juan de Dios Hospital.
  This programme is divided into 5 phases, each of these phases coincides with a level of the gait assessment scale. Each individual will start at the level assigned by the doctor and will only have access to the videos of the indicated level and the levels below it. As the patient meets the recovery goals, the physician will provide access to the higher level videos.The functional recovery plan begins the day after the hip fracture and continues after the patient has been discharged for a total of 16 weeks.
  Groups: Non-exposed cohort (protective factor)
Other: Standardised nursing care plan — Consisting of postural changes described in the standardised nursing care plan. Within this plan, the patient was moved to a sitting position prematurely (within the first 24 hours) and started to ambulate within the following 48 hours, provided that the patient's general condition allowed it. This group did not receive any specific functional recovery plan.
  Groups: Exposed cohort (retrospective)

SUMMARY:
Background In recent years, Western populations have experienced an increase in life expectancy and therefore an ageing population. This has led to an increase in the number of low-energy hip fractures, which have a major impact in terms of mortality, mobility and loss of function in activities of daily living in this segment of the population.

Objectives To determine the impact in terms of functional recovery, return to pre-hip fracture functional status, of elderly patients treated with the new multimodal therapeutic exercise programme and follow-up for one year compared to patients treated with the previously developed standardised nursing care plan at the Hospital San Juan de Dios de León.

Methodology Ambispective observational study of cohort with two groups, an exposed cohort (retrospective) and a non-exposed cohort (protective factor), made up of people over 65 years of age referred from the Emergency Department of the University Care Centre of León (CAULE) with a confirmed diagnosis of hip fracture, who underwent hip fracture surgery in theHospital San Juan de Dios de León during the years 2020 and 2021.

In order to carry out an analysis of the new care model proposed by the area of orthogeriatrics for the year 2021: functional recovery programme and its follow-up through a digital application, the entire simple universe will be included (analysis of the complete cohort) with follow-up over a period of one year.

DETAILED DESCRIPTION:
This research project is intended to be carried out in the Functional Recovery Unit integrated in the Orthogeriatrics Service of the San Juan de Dios Hospital and has the following work plan:

* Administrative Phase. Complete development of the project in writing and submission for approval to the Doctoral Commission of the University of Murcia and the Research Commission of the Order of San Juan de Dios. Once the project has been approved, it will be submitted to the Clinical Research Ethics Committee (CEIC) as deemed appropriate.
* Initial Phase-Start-up. Duration 18 months. The programme will start when the patient is admitted to hospital for hip fracture. Participants who meet the eligibility criteria for the study will be recruited and data collected participants will be informed of the purpose of the study and their written informed consent will be requested.

Description of the process:

* Candidate selection: the patient will be cared for by orthogeriatrics unit according to its standard clinical practice protocol approved by the medical management, and based on the care model established by the National Hip Fracture Registry.
* If the patient is admitted from the emergency department, a referral to geriatrics will be requested to assess the patient.
* Explanation of the programme and request for informed consent: at the time of admission, an interview will be held between the patient or relative and the doctor in charge (traumatology service) explaining the process for patients with osteoporotic hip fracture in the Hospital; which encompasses the set of coordinated medical decisions (Emergency, Traumatology, Geriatrics) with the aim of obtaining the highest quality care, shorter hospital stay with the maximum level of independence and avoiding a second fracture. In the same way and at the same time, the multimodal plan of therapeutic exercise and functional recovery that will help them during their recovery process will be explained to them.

Subsequently, the patient will be informed of the data collection process, mobile application and follow-up for 1 year, and signatures will be requested for informed consent for anaesthesia, surgery and participation in the study.

Profiles of patients whose clinical circumstances permit, a corroborated history should be taken, including:

* Premorbid function and mobility.
* Available social support (including whether the patient already has a caregiver or whether someone is willing and able to provide such support)
* Relevant current clinical conditions
* State of mind.

  * Hip Surgery.
  * Recovery programme (protocol of action that replaces the usual practice developed previously):
* Specific hip fracture recovery programme,restoring the mobility, strength and balance of the operated patient, in order to facilitate the return to a functional state as close as possible to the state prior to surgery and in the shortest possible time. This programme is part of the standard treatment protocol implemented since January 2021 by the Orthogeriatrics Unit of the San Juan de Dios Hospital.

This programme is divided into 5 phases, each of these phases coincides with a level of the gait assessment scale. Each individual will start at the level assigned by the doctor and will only have access to the videos of the indicated level and the levels below it. As the patient meets the recovery goals, the physician will provide access to the higher level videos.The functional recovery plan begins the day after the hip fracture and continues after the patient has been discharged for a total of 16 weeks.

o The therapeutic plan for the historical control group (standard practice until 31 December 2020) consisting of postural changes described in the standardised nursing care plan. Within this plan, the patient was moved to a sitting position prematurely (within the first 24 hours) and started to ambulate within the following 48 hours, provided that the patient's general condition allowed it. This group did not receive any specific functional recovery plan.

* The patient is discharged from hospital and will be assigned a link where he/she will be able to access the online platform to send information from the questionnaires sent during the established periods of 1, 3, 6 and 12 months and will also be sent videos illustrating the rehabilitation exercises that he/she will have to perform during this period. The patient and/or carer will be explained how the tool works, how to access the digital information content and how to access the questionnaires. A means of contact will be provided to resolve doubts, if any. The PI will have access through the web/app platform to a control panel where he/she will be able to detect a patient's lack of adherence, if any, or alerts related to clinical evolution, allowing for exhaustive monitoring of the patient.
* Analysis of results: The data collected will be analysed with the Statistical Package for the Social Sciences programme. The mean, median and standard deviation of each of the variables will be calculated. Based on the data obtained from the existing literature, having selected a sample of 67 patients, a normal distribution can be assumed for all variables For baseline demographic and clinical characteristics, a comparison of means for quantitative variables (t-Student), and of proportions (Chi-square) for qualitative will be performed The statistical analysis will be carried out with a confidence level of 95%, so that statistically significant values will be considered to be those whose probability is < 0.05.
* Dissemination of results: the results of this study will be presented for dissemination in scientific journals and specialised conferences.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred from the Emergency Service of the León Assistance Complex (CAULE), confirmation of the medical diagnosis of hip fracture by means of Antero-Posterior and Lateral radiography.
* Be over 65 years of age.
* Be able to walk before the fracture with or without the help of instruments or people.
* Have signed the informed consent to participate in the research project.
* With access to a mobile phone with the option to install applications.

Exclusion Criteria:

* Multiple trauma patients will be excluded.
* Metastatic origin of the fracture.
* Periprosthetic fracture.
* Patients with cognitive impairment that makes it impossible for them to use a mobile phone with applications and who are not accompanied by a responsible person during the recovery process.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The target population will be made up of people over 65 years of age referred from the Emergency Department of the Centro Asistencial Universitario de León (CAULE) with a confirmed diagnosis of hip fracture, who are going to undergo hip fracture surgery at the HSJD.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-21 (Estimated); Study Completion 2022-08-21 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Classification-1d. | First day
  Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
  Level 0: Patient who cannot remain seated for more than 1 minute without the help of the backrest and the armrest.
  Level 1: Patient who can remain seated without the help of the backrest and the armrest for more than 1 minute.
  Level 2: non-functional ambulation. Walking with great physical assistance. Level 3: home walking, walking with light physical contact with a person. Level 4: walks autonomously in the environment of the house or neighborhood, but needs supervision of a person.
  Level 5: independent community wandering.
Functional Ambulation Classification-3dQX. | 3 days after surgery
  Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
  Level 0: Patient who cannot remain seated for more than 1 minute without the help of the backrest and the armrest.
  Level 1: Patient who can remain seated without the help of the backrest and the armrest for more than 1 minute.
  Level 2: non-functional ambulation. Walking with great physical assistance. Level 3: home walking, walking with light physical contact with a person. Level 4: walks autonomously in the environment of the house or neighborhood, but needs supervision of a person.
  Level 5: independent community wandering.
Functional Ambulation Classification-6W. | 6 weeks
  Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
  Level 0: Patient who cannot remain seated for more than 1 minute without the help of the backrest and the armrest.
  Level 1: Patient who can remain seated without the help of the backrest and the armrest for more than 1 minute.
  Level 2: non-functional ambulation. Walking with great physical assistance. Level 3: home walking, walking with light physical contact with a person. Level 4: walks autonomously in the environment of the house or neighborhood, but needs supervision of a person.
  Level 5: independent community wandering.
Functional Ambulation Classification-16W. | 16 weeks
  Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
  Level 0: Patient who cannot remain seated for more than 1 minute without the help of the backrest and the armrest.
  Level 1: Patient who can remain seated without the help of the backrest and the armrest for more than 1 minute.
  Level 2: non-functional ambulation. Walking with great physical assistance. Level 3: home walking, walking with light physical contact with a person. Level 4: walks autonomously in the environment of the house or neighborhood, but needs supervision of a person.
  Level 5: independent community wandering.
Functional Ambulation Classification-1Y. | 1 year
  Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
  Level 0: Patient who cannot remain seated for more than 1 minute without the help of the backrest and the armrest.
  Level 1: Patient who can remain seated without the help of the backrest and the armrest for more than 1 minute.
  Level 2: non-functional ambulation. Walking with great physical assistance. Level 3: home walking, walking with light physical contact with a person. Level 4: walks autonomously in the environment of the house or neighborhood, but needs supervision of a person.
  Level 5: independent community wandering.

SECONDARY OUTCOMES:
Short Portable Mental Status Questionnaire 1d | First day
  Evaluates the cognitive state of the patient at the time of administration. It consists of 10 questions that are asked prior to the surgical intervention, in which errors are computed. It is proposed to perform the test at the time closest to the baseline cognitive situation of the patient.
  What day is today? (Month, day, Year). What day of the week is today? Where are we now? What is your phone number? (If there is no phone, street address). How old are you? What is your date of birth? Who is the current Prime Minister? Who was the previous Prime Minister? Tell me the first surname of his mother. Starting at 20, subtract from 3 to 3 successively until you reach 0.
Short Portable Mental Status Questionnaire 3dQx | 3 days after surgery
  Evaluates the cognitive state of the patient at the time of administration. It consists of 10 questions that are asked prior to the surgical intervention, in which errors are computed. It is proposed to perform the test at the time closest to the baseline cognitive situation of the patient.
  What day is today? (Month, day, Year). What day of the week is today? Where are we now? What is your phone number? (If there is no phone, street address). How old are you? What is your date of birth? Who is the current Prime Minister? Who was the previous Prime Minister? Tell me the first surname of his mother. Starting at 20, subtract from 3 to 3 successively until you reach 0.
Mobility prior to the fracture, according to the Spanish national registry of hip fractures due to fragility 1d. | First day
  It evaluates by levels of capacity that range between 0 and 11. Its design allows to determine first the capacity of the gait and, secondly, to see the evolution and establish treatment guidelines.
Mobility prior to the fracture, according to the Spanish national registry of hip fractures due to fragility 3dQx. | 3 days after surgery
  It evaluates by levels of capacity that range between 0 and 11. Its design allows to determine first the capacity of the gait and, secondly, to see the evolution and establish treatment guidelines.
Mobility prior to the fracture, according to the Spanish national registry of hip fractures due to fragility 6W. | 6 weeks
  It evaluates by levels of capacity that range between 0 and 11. Its design allows to determine first the capacity of the gait and, secondly, to see the evolution and establish treatment guidelines.
Mobility prior to the fracture, according to the Spanish national registry of hip fractures due to fragility 16W. | 16 weeks
  It evaluates by levels of capacity that range between 0 and 11. Its design allows to determine first the capacity of the gait and, secondly, to see the evolution and establish treatment guidelines.
Mobility prior to the fracture, according to the Spanish national registry of hip fractures due to fragility 1Y. | 1 year
  It evaluates by levels of capacity that range between 0 and 11. Its design allows to determine first the capacity of the gait and, secondly, to see the evolution and establish treatment guidelines.
Barthel Index 1d. | First day
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living. Each performance item is rated on this scale with a given number of points assigned to each level or ranking:
  Values: 0-20 total dependency. Values: 21-60 severe dependency. Values: 61-90 moderate dependence. Values: 91-99 low dependency Values: 100 independence.
Barthel Index 3dQx | 3 days after surgery
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living. Each performance item is rated on this scale with a given number of points assigned to each level or ranking:
  Values: 0-20 total dependency. Values: 21-60 severe dependency. Values: 61-90 moderate dependence. Values: 91-99 low dependency Values: 100 independence.
Barthel Index 6W | 6 weeks
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living. Each performance item is rated on this scale with a given number of points assigned to each level or ranking:
  Values: 0-20 total dependency. Values: 21-60 severe dependency. Values: 61-90 moderate dependence. Values: 91-99 low dependency Values: 100 independence.
Barthel Index 16W | 16 weeks
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living. Each performance item is rated on this scale with a given number of points assigned to each level or ranking:
  Values: 0-20 total dependency. Values: 21-60 severe dependency. Values: 61-90 moderate dependence. Values: 91-99 low dependency Values: 100 independence.
Barthel Index 1Y | 1 year
  The Barthel scale is an ordinal scale used to measure performance in activities of daily living. Each performance item is rated on this scale with a given number of points assigned to each level or ranking:
  Values: 0-20 total dependency. Values: 21-60 severe dependency. Values: 61-90 moderate dependence. Values: 91-99 low dependency Values: 100 independence.
SARC-F questionnaire (Sarcopenia Screening) 1d | First day
  SARC-F is a simple questionnaire to rapidly diagnose of sarcopenia. The maximum score is 10 points. If after the test the score is <4 points indicates an acceptable state of health, while any score higher than the previous one indicates risk of sarcopenia.
SARC-F questionnaire (Sarcopenia Screening) 3dQx | 3 days after surgery
  SARC-F is a simple questionnaire to rapidly diagnose of sarcopenia. The maximum score is 10 points. If after the test the score is <4 points indicates an acceptable state of health, while any score higher than the previous one indicates risk of sarcopenia.
SARC-F questionnaire (Sarcopenia Screening) 6W | 6 weeks
  SARC-F is a simple questionnaire to rapidly diagnose of sarcopenia. The maximum score is 10 points. If after the test the score is <4 points indicates an acceptable state of health, while any score higher than the previous one indicates risk of sarcopenia.
SARC-F questionnaire (Sarcopenia Screening) 16W | 16 weeks
  SARC-F is a simple questionnaire to rapidly diagnose of sarcopenia. The maximum score is 10 points. If after the test the score is <4 points indicates an acceptable state of health, while any score higher than the previous one indicates risk of sarcopenia.
SARC-F questionnaire (Sarcopenia Screening) 1Y | 1 year
  SARC-F is a simple questionnaire to rapidly diagnose of sarcopenia. The maximum score is 10 points. If after the test the score is <4 points indicates an acceptable state of health, while any score higher than the previous one indicates risk of sarcopenia.
Oxford Hip Score 1d | First day
  The Oxford Hip Score is a patient-centered questionnaire that is designed to assess functional ability and pain from the patient's perspective. It is a short, twelve-item questionnaire developed for completion by patients undergoing surgery and is extensively referenced in the orthopedic literature.
  Results:
  0-19: Severe impact. 20-29: Moderate to severe impact. 30-39: Mild to moderate impact. 40-48: Satisfactory condition.
Oxford Hip Score 3dQx | 3 days after surgery
  The Oxford Hip Score is a patient-centered questionnaire that is designed to assess functional ability and pain from the patient's perspective. It is a short, twelve-item questionnaire developed for completion by patients undergoing surgery and is extensively referenced in the orthopedic literature.
  Results:
  0-19: Severe impact. 20-29: Moderate to severe impact. 30-39: Mild to moderate impact. 40-48: Satisfactory condition.
Oxford Hip Score 6W | 6 weeks
  The Oxford Hip Score is a patient-centered questionnaire that is designed to assess functional ability and pain from the patient's perspective. It is a short, twelve-item questionnaire developed for completion by patients undergoing surgery and is extensively referenced in the orthopedic literature.
  Results:
  0-19: Severe impact. 20-29: Moderate to severe impact. 30-39: Mild to moderate impact. 40-48: Satisfactory condition.
Oxford Hip Score 16W | 16 weeks
  The Oxford Hip Score is a patient-centered questionnaire that is designed to assess functional ability and pain from the patient's perspective. It is a short, twelve-item questionnaire developed for completion by patients undergoing surgery and is extensively referenced in the orthopedic literature.
  Results:
  0-19: Severe impact. 20-29: Moderate to severe impact. 30-39: Mild to moderate impact. 40-48: Satisfactory condition.
Oxford Hip Score 1Y | 1 year
  The Oxford Hip Score is a patient-centered questionnaire that is designed to assess functional ability and pain from the patient's perspective. It is a short, twelve-item questionnaire developed for completion by patients undergoing surgery and is extensively referenced in the orthopedic literature.
  Results:
  0-19: Severe impact. 20-29: Moderate to severe impact. 30-39: Mild to moderate impact. 40-48: Satisfactory condition.
STRATIFY 1d. | First day
  The STRATIFY score range from 0 to 5 points and the predictive cut off of risk of falling. The total score of the STRATIFY scale is obtained based on the sum of the answers referring to the five questions, being able to take values between zero and five. A score of 0 corresponds to a risk considered low, equal to 1 corresponds to a moderate risk and, finally, greater than or equal to 2 corresponds to a high risk
STRATIFY 3dQx | 3 days after surgery
  The STRATIFY score range from 0 to 5 points and the predictive cut off of risk of falling. The total score of the STRATIFY scale is obtained based on the sum of the answers referring to the five questions, being able to take values between zero and five. A score of 0 corresponds to a risk considered low, equal to 1 corresponds to a moderate risk and, finally, greater than or equal to 2 corresponds to a high risk
STRATIFY 6W | 6 weeks
  The STRATIFY score range from 0 to 5 points and the predictive cut off of risk of falling. The total score of the STRATIFY scale is obtained based on the sum of the answers referring to the five questions, being able to take values between zero and five. A score of 0 corresponds to a risk considered low, equal to 1 corresponds to a moderate risk and, finally, greater than or equal to 2 corresponds to a high risk
STRATIFY 16W | 16 weeks
  The STRATIFY score range from 0 to 5 points and the predictive cut off of risk of falling. The total score of the STRATIFY scale is obtained based on the sum of the answers referring to the five questions, being able to take values between zero and five. A score of 0 corresponds to a risk considered low, equal to 1 corresponds to a moderate risk and, finally, greater than or equal to 2 corresponds to a high risk
STRATIFY 1Y | 1 year
  The STRATIFY score range from 0 to 5 points and the predictive cut off of risk of falling. The total score of the STRATIFY scale is obtained based on the sum of the answers referring to the five questions, being able to take values between zero and five. A score of 0 corresponds to a risk considered low, equal to 1 corresponds to a moderate risk and, finally, greater than or equal to 2 corresponds to a high risk

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Zambrano Martín, MSC PT, Principal Investigator — Centro Universitario San Rafael
Locations (1):
- Hospital San Juan de Dios de León, León, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT04919083/Prot_SAP_ICF_000.pdf